CLINICAL TRIAL: NCT06171841
Title: Acute and Chronic Effects of Low-Intensity Blood Flow Restriction Training in Normoxia and Hypoxia Conditions on Muscle Strength, Thickness, Catecholamine, and Inflammatory Responses in Physically Active Adults
Brief Title: Effects of Low-Intensity Blood Flow Restriction Training in Normoxia and Hypoxia Conditions
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Jerzy Kukuczka Academy of Physical Education in Katowice (Other)
Responsible Party: Principal Investigator, Michal Krzysztofik, Associate Professor, The Jerzy Kukuczka Academy of Physical Education in Katowice
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SKN/SP/569582/2023
Record Dates: First submitted 2023-11-25; First posted 2023-12-15 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Hypoxia, Altitude; Blood Flow Restriction; Resistance Training
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Low-Intensity Normoxia (Active Comparator): Participants will be breathing room air, and perform low-intensity lower-body resistance exercise.
  Interventions: Other: low-intensity resistance training
- High-Intensity Normoxia (Active Comparator): Participants will be breathing room air, and perform high-intensity lower-body resistance exercise.
  Interventions: Other: high-intensity resistance training
- Low-Intensity Normoxia with Blood Flow Restriction (Experimental): Participants will be breathing room air, and perform low-intensity lower-body resistance exercise combined with blood flow restriction.
  Interventions: Other: low-intensity resistance training combined with blood flow restriction
- Low-Intensity Hypoxia (Experimental): Participants will be breathing a 13% oxygen gas mixture, and perform low-intensity lower-body resistance exercise.
  Interventions: Other: low-intensity resistance training in hypoxia condition
- Low-Intensity Hypoxia with Blood Flow Restriction (Experimental): Participants will be breathing a 13% oxygen gas mixture, and perform low-intensity lower-body resistance exercise combined with blood flow restriction.
  Interventions: Other: low-intensity resistance training combined with blood flow restriction in hypoxia condition

INTERVENTIONS:
Other: low-intensity resistance training — 4 sets of 30/15/15/15 repetitions of leg press exercise with a load of 20-30% of one-repetition maximum (weeks 1-3: 20%, weeks 4-6: 30%) in normoxic conditions performed twice a week for 6 weeks.
  Arms: Low-Intensity Normoxia
Other: high-intensity resistance training — 4 sets of 10 repetitions of leg press exercise at 70-80% one-repetition maximum (weeks 1-3: 70%, weeks 4-6: 80%) in normoxic conditions performed twice a week for 6 weeks.
  Arms: High-Intensity Normoxia
Other: low-intensity resistance training combined with blood flow restriction — 4 sets of 30/15/15/15 repetitions of leg press exercise with a load of 20-30% of one-repetition maximum (weeks 1-3: 20%, weeks 4-6: 30%) in normoxic conditions with lower-limbs blood flow restriction (80% total occlusion pressure) performed twice a week for 6 weeks.
  Arms: Low-Intensity Normoxia with Blood Flow Restriction
Other: low-intensity resistance training in hypoxia condition — 4 sets of 30/15/15/15 repetitions of leg press exercise with a load of 20-30% of one-repetition maximum (weeks 1-3: 20%, weeks 4-6: 30%) in hypoxia conditions (3500 meters above sea) performed twice a week for 6 weeks.
  Arms: Low-Intensity Hypoxia
Other: low-intensity resistance training combined with blood flow restriction in hypoxia condition — 4 sets of 30/15/15/15 repetitions of leg press exercise with a load of 20-30% of one-repetition maximum (weeks 1-3: 20%, weeks 4-6: 30%) in normobaric hypoxia conditions (3500 meters above sea) with lower-limbs blood flow restriction (80% total occlusion pressure) performed twice a week for 6 weeks.
  Arms: Low-Intensity Hypoxia with Blood Flow Restriction

SUMMARY:
One approach to significantly reducing resistance training intensity while maintaining effectiveness in muscle mass and strength development involves conducting training sessions under hypoxic conditions. This is likely due to heightened physiological responses. While sports science research indicates a substantial impact of hypoxic conditions on immediate increases in metabolic stress and augmented hormonal responses, recent findings suggest that the role of their influence on skeletal muscle adaptations post-resistance training under hypoxic conditions remains unknown. Additionally, there is a lack of reports on whether the type of hypoxia applied via blood flow restriction or chamber differentiates the increase in secretion of these catecholamines in both immediate and long-term aspects.

ELIGIBILITY:
Inclusion Criteria:

* Regularly physically active (at least 30 mins of structured exercise 3 times per week),
* Sea-level natives,
* Experienced in resistance training (at least one year of experience in regular resistance exercise)

Exclusion Criteria:

* presence of any medical risk factors to exercise and/or exposure to altitude
* presence of any medical condition that would make the protocol unreasonably hazardous for the participant
* smokers

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-06-20 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Force Output | Immediately pre and post first and last training session
  Force plate will be used to quantify maximum absolute (N) and relative force output (body mass divided per force output in N/kg) during maximum voluntary isometric back squat in a 100ms time frame. Participants will be pushing as hard and as fast as they can on an unmoveable barbell while standing on a force plate.
One-Repetition Maximum | within 5 days from the start and end of training
  One-Repetition Maximum test in leg press exercise will be performed to quantify maximum lower body dynamic strength (kg). Participants will be performing single repetitions of leg press exercise with increasing load until volitional failure.
Maximum Number of Repetitions | within 5 days from the start and end of training
  A maximum number of repetitions in leg press exercise will be performed to quantify lower body strength endurance (number). Participants will be performing leg press exercise at 50% of one-repetition maximum until volitional failure.
Countermovement Jump Height | Immediately pre and post first and last training session
  Countermovement jump height will be performed estimated via take-off velocity performed on force plates to Participants will perform 3 trials on force plate.
Countermovement Jump Power Output | Immediately pre and post first and last training session
  Countermovement jump performance will be performed to quantify maximum lower body relative and absolute power-output (W/kg and W), and jump height (cm) with concomitant assessment of contraction depth (cm) and contraction time (ms). Participants will perform 3 trials on force plate.
Catecholamine Response | Immediately pre and post first and last training session
  A blood sample will be analyzed to quantify changes in epinephrine and norepinephrine level changes.
Muscle Stiffness | Immediately pre and post first and last training session
  Myotonometry measure will be used to quantify changes in vastus medialis oblique muscle stiffness in N/m
Muscle Thickness | within 5 days from the start and end of training
  Ultrasonography measure will be used to quantify changes in vastus medialis oblique cross-sectional area.

SECONDARY OUTCOMES:
Perception of Pain | Immediately pre and post every training session
  A visual analogue scale will be used to quantify the perception of pain (units on a scale).
Perception of Effort | Immediately pre and post every training session
  The rate of perceived exertion scale will be used to quantify the perception of effort (units on a scale).
Blood Pressure | Immediately pre and post first and last training session
  Systolic and diastolic blood pressure will be measured to quantify blood pressure responses.

OTHER OUTCOMES:
Total Body Mass | within 5 days from the start and end of training
  Dual-energy X-ray absorptiometry will be used to quantify total body mass (kg).
Percentage Body Fat | within 5 days from the start and end of training
  Dual-energy X-ray absorptiometry will be used to quantify the percentage of body fat (%).
Bone Mass Density | within 5 days from the start and end of training
  Dual-energy X-ray absorptiometry will be used to quantify femur bone mass density (g/cm2).
Bone Mineral Content | within 5 days from the start and end of training
  Dual-energy X-ray absorptiometry will be used to quantify bone mineral content (g).

CONTACTS AND LOCATIONS:
Locations (1):
- The Jerzy Kukuczka Academy of Physical Education, Katowice, Silesian Voivodeship, Poland